CLINICAL TRIAL: NCT05451290
Title: Camrelizumab Plus Apatinib Combined With GEMOX (Gemcitabine and Oxaliplatin ) in the Perioperative Treatment of Locally Advanced Biliary Tract Malignancies: A Prospective, Multicenter, Phase Ⅱ Study
Brief Title: Camrelizumab Plus Apatinib in Combination With GEMOX (Gemcitabine and Oxaliplatin ) in Patients With Locally Advanced Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220057C
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Biliary Tract Carcinoma
MeSH Terms: interventions — camrelizumab; apatinib; Gemcitabine; Oxaliplatin; Tegafur; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Camrelizumab, apatinib, gemcitabine, oxaliplatin, tegafur

INTERVENTIONS:
Drug: Camrelizumab, apatinib, gemcitabine, oxaliplatin, tegafur — Perioperative treatment: camrelizumab plus apatinib in combination with GEMOX 2-4 cycles (neoadjuvant); camrelizumab plus S-1 up to 1 year (adjuvant).
  Other Names: surgery

SUMMARY:
This is a phase II open-label, one-arm, multicenter study aimed to explore the efficacy and safety of perioperative (neoadjuvant and adjuvant) treatment for patients with advanced biliary tract carcinoma.

DETAILED DESCRIPTION:
Enrolled participants should be treated with neoadjuvant camrelizumab and apatinib and GEMOX, after surgery, be treated with adjuvant camrelizumab and S-1.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent document must be signed.
2. Aged 18-75 years old, both genders.
3. Pathologically confirmed biliary tract adenocarcinoma and haven't been treated before.
4. An Eastern Cooperative Oncology Group performance status of 0 to 1.
5. Locally advanced biliary tract adenocarcinoma confirmed by MDT discussion.
6. The function of vital organs meets the following requirements:

   the blood ANC count≥1.5x109 /L; hemoglobin ≥ 90 g/L，the blood platelet count≥80 x109 /L, total bilirubin ≤ 1.5 x ULN, ALT and AST ≤3 x ULN(< 5 x ULN for patients with live metastasis), serum creatinine≤1.5 x ULN, endogenous creatinine clearance rate ≥45ml/min.
7. At least 1 measurable lesion as defined by RECIST 1.1.
8. Women of reproductive age need to take effective contraceptive measures during and within 3 months of the end of medication.
9. Subjects should have good compliance and cooperate with the follow-up.

Exclusion Criteria:

1. Subject has any active autoimmune disease or history of autoimmune disease will not be included, nor will patients with active tuberculosis or hepatitis or HIV.
2. Subjects with illness or medical conditions that could jeopardize their sugery, such as severe cardiopulmonary insufficiency and coagulation disorders, cannot be enrolled.
3. Subjects with active malignancies other than BTC within 5 years should be excluded, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix and superficial bladder cancer [Ta, Tis & T1] and papillary thyroid cancer.
4. Any unstable systemic disease which might need systemic treatment should not be enrolled (including active infection, liver or renal disease, metabolic disease, acute cerebral infarction or hemorrhage), or serious co-morbidities that by the judgment of the investigator, may compromise the patient's safety or impair the patient's ability to complete the study.
5. Subjects who have significant cardiovascular events should not be enrolled, for example: congestive heart failure > NYHA class 2, unstable angina, active coronary artery disease (CAD) (only allow the subjects with presence of myocardial infarction more than 1 year prior to study); severe arrhythmias in need of treatment (only allow those been treated with β-blockers or digoxin) or uncontrolled hypertension.
6. Subjects with history of neurological or psychiatric disease, including epilepsy or dementia or diseases alike should not be enrolled.
7. Subjects with interstitial lung disease or a history of interstitial pneumonia should not be enrolled.
8. Subjects who had participated in other anti-tumor clinical trials within 4 weeks prior to enrollment should be avoided.
9. Subjects who had used PD-1/PD-L1 or other antitumor immunotherapeutic agents prior to enrollment should be avoided.
10. The following subjects should be avoided: pregnant or lactating women; those who have childbearing potential and unwilling or unable to use effective contraception measures.
11. Other circumstances that could affect the trial or the result of the study judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
1-year EFS rate | 1 year
  EFS was defined as the time from the first administration of study treatment to the first occurrence of any of the following events: disease progression that precluded surgical resection, disease recurrence after curative-intent surgery, disease progression in patients who did not undergo surgery, or death from any cause. 1-year EFS rate was the incidence rate of event-free survival within one year.

SECONDARY OUTCOMES:
R0 resection rate | up to 2 years
  The proportion of patients who underwent complete tumor resection with microscopically negative margins
Major pathologic response (MPR) | up to 2 years
  10% or less residual viable tumor cells in the resected specimen
ORR | up to 2 years
  The proportion of patients with a confirmed complete or partial response
DCR | up to 2 years
  The proportion of patients with a complete response, partial response, or stable disease
EFS | up to 5 years
  EFS was defined as the time from the first administration of study treatment to the first occurrence of any of the following events: disease progression that precluded surgical resection, disease recurrence after curative-intent surgery, disease progression in patients who did not undergo surgery, or death from any cause.
OS | up to 5 years
  The time from the first dose of study treatment to death from any cause
adverse event | up to 2 years
  Based on the assessment using CTCAE v5.0, the safety was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No